CLINICAL TRIAL: NCT01509196
Title: Open-label, Randomized Comparative Study to Evaluate the Pharmacokinetic Characteristics of Fenofibric Acid Between Lipidilsupra Tablet and HIP0901 Capsule in Healthy Male Subjects
Brief Title: A Bioequivalence Study Comparing HIP0901 Capsule With Lipidilsupra Tablet
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-FEN-101
Record Dates: First submitted 2012-01-10; First posted 2012-01-12 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Healthy
Keywords: Fenofibric acid; HIP0901; Lipidilsupra

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HIP0901 (Experimental): Fenofibric acid
  Interventions: Drug: HIP0901 / Lipidilsupra
- Lipidilsupra (Active Comparator): Fenofibrate
  Interventions: Drug: HIP0901 / Lipidilsupra

INTERVENTIONS:
Drug: HIP0901 / Lipidilsupra — HIP0901 capsule(Fenofibric acid, 135mg) / Lipidilsupra tablet(Fenofibrate, 160mg)

SUMMARY:
The purpose of this study is to evaluate pharmacokinetics and safety after oral administration of HIP0901 capsules and Lipidilsupra tablets.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age between 20 and 45
* Informed of the investigational nature of this study and voluntarily agree to participate in this study
* Weight>50kg, BMI of >18kg/m2 and <27kg/m2 subject

Exclusion Criteria:

* Acute disease within 28 days prior to start of study drug administration
* Use of any prescription medication within 14 days prior to Day 1
* Use of any medication within 7 days prior to Day 1
* Has a severe medical history of hypersensitivity to fibric acid derivative
* Participation in another clinical study within 30 days prior to start of study drug administration

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
AUC of Fenofibric acid | 0-96 hrs
Cmax of Fenofibric acid | 0-96 hrs

CONTACTS AND LOCATIONS:
Overall Officials: Ji-Young Park, MD, PhD, Principal Investigator — Korea University Anam Hospital
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea